CLINICAL TRIAL: NCT06586086
Title: The Effect of Anxiety on Pain-pressure Threshold in a Healthy Population
Status: Suspended | Type: Observational
Why Stopped: On hold pending challenges in scheduling for PI
Sponsor: Philadelphia College of Osteopathic Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 082419
Record Dates: First submitted 2024-08-16; First posted 2024-09-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study recruit individuals who are 18 years of age AND Do NOT have a history of diagnosed anxiety disorders AND Do NOT currently have any area of pain lasting 3 months or longer.

The study will measure discomfort with a controlled application of pressure to different muscles and compare these measures with the individual's score on a standardized assessment of anxiety.

DETAILED DESCRIPTION:
Purpose Anxiety in general has been associated with lower (more sensitive) pain-pressure thresholds, however, to the best of the investigators knowledge, no research has attempted to differentiate state versus trait anxiety and their respective impacts on pressure sensitivity.

Trait anxiety is an individuals tendency to appraise situations as threatening, avoid anxiety provoking situations, and demonstrate high baseline physiological arousal. State anxiety is defined as; transient state of arousal subjectively experienced as anxiety; This study's objective is to differentiate the role of each anxiety subscale in systemic sensory perception changes. This data may better allow clinicians to glean accurate data about an individuals baseline symptoms as well as potentially shedding light on state-related changes in pain thresholds.

Objectives The primary objective of this study will be to elucidate the differing relationships of trait anxiety and state anxiety on pain-pressure threshold (PPT.) While other measures exist to gauge potential sensitization to sensory stimuli, PPT is often chosen for research due to the ease of administration and its ability to translate data into practice.

Study Population Target population will be healthy adults age 18+. As will be delineated further in this document, this study will recruit healthy adults such as to minimize potential modifications in sensory perception due to comorbidities, medication etc.

Number of Participants The study will enroll 60 participants to provide more robust statistical power

Study Design The study will be a descriptive, cross-sectional design. The study will seek to draw associations between the different anxiety subscales and the subject's pain-pressure threshold. No variables will be manipulated.

Study Duration The study participants will complete the STAI-5, a validated short version of the State-Trait Anxiety Inventory. Immediately after questionnaire administration participants will be tested for pain-pressure thresholds. Each participant session will last approximately 30 minutes. The entire study duration will be 20 weeks to allow for test administration for all participants.

Outcome Variables The outcome variable in question is pain-pressure threshold for the bilateral upper trapezius, extensor carpi radialis, Tibialis anterior, and lumbar paraspinal (L3 segment level) muscles. Each site will be tested three times, and the results will be averaged. The mean score from both sides will also subsequently be averaged to provide a single numerical outcome for each participant. PPT data for each participant will be compared with both Trait and State anxiety scores from the STAI-5 tool.

Locations/Facilities The research will be conducted entirely within the research suite in the Physical Therapy Department of the Philadelphia College of Osteopathic Medicine-Georgia Campus, Suwanee, GA.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Able to read and complete the STAI-5 questionnaire as written in English

Exclusion Criteria:

* Pain lasting three months or longer, located anywhere in the body
* Severe health problem (such as cancer, cardiac, neurologic or psychiatric/anxiety disorders),
* Current pregnancy and/or gave birth in the last year.
* Subjects currently taking medication which may impact sensory processing, such as antidepressants, opioids, neuroleptics, anticonvulsive drugs or steroids.
* Subjects diagnosed with fibromyalgia or other conditions known to reduce muscular pain-pressure thresholds, such as Lyme disease, polymyalgia, Lupus and Rheumatoid Arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain-Pressure Threshold | A single collection session of data for each participant, lasting approximately 30 minutes, performed after completion of the STAI-5. Total Data collection window is 4 months.
  Quantitative measurement of the amount of pressure applied at the point when the subject described the pressure as slight discomfort

SECONDARY OUTCOMES:
State-Trait Anxiety questionnaire (STAI)-5 question form | A single collection session of data for each participant, lasting approximately 5 minutes. Total Data collection window is 4 months
  A standardized test which measures both state and trait anxiety. Consists of two subscales, trait anxiety and state anxiety. Each section score ranges from 5 to 20, with a higher score indicating higher anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lowe, Principal Investigator — PCOM GA
Locations (1):
- Philadelphia College of Osteopathic Medicine-Georgia Campus, Suwanee, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pending requirements of potential publication avenues